CLINICAL TRIAL: NCT04000685
Title: The Effects of Different Exercise Approaches on Physical and Cognitive Variables in Patients With Chronic Low Back Pain
Brief Title: The Effects of Different Exercise Approaches in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Muzeyyen Oz, Research Assistant, Neck and Low Back Health Unit, Principal Investigator, MSc, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-19029
Record Dates: First submitted 2019-06-23; First posted 2019-06-27 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Chronic Low-back Pain
Keywords: low back pain; exercise; cognitive; aerobic; yoga
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga exercise group (Active Comparator): Yoga program were applied all patients in this group accompanied by physiotherapist. Sessions included selected breathing, warm up and relaxation exercises.
  Interventions: Other: Yoga exercise program
- Spinal stabilization exercise group (Active Comparator): Spinal stabilization exercise with three different progressive phases were applied all patients in this group accompanied by physiotherapist.
  Interventions: Other: Spinal stabilization exercise program
- aerobic walking exercise group (Active Comparator): Aerobic walking exercise program applied all patients in this group accompanied by physiotherapist.
  Interventions: Other: Aerobic walking program

INTERVENTIONS:
Other: Yoga exercise program — Yoga exercise program will be applied two sessions per week, totally eight week.
  Arms: Yoga exercise group
Other: Spinal stabilization exercise program — Spinal stabilization exercise program will be applied two sessions per week, totally eight week.
  Arms: Spinal stabilization exercise group
Other: Aerobic walking program — Aerobic walking program will be applied two sessions per week, totally eight week.
  Arms: aerobic walking exercise group

SUMMARY:
Identification of the effects of yoga, stabilization exercise and aerobic exercise approaches on physical and cognitive variables in individuals with low back pain.

DETAILED DESCRIPTION:
Patients participating in the study were divided three parallel groups. The patients in the stabilization exercise group were instructed to perform spinal stabilization exercises, the patients in the yoga group were instructed to perform yoga program consisting of breathing, relaxation and flexibility exercises. The patients in the aerobic exercise group were instructed to perform aerobic walking training. The severity of the pain evaluated through visual analog scale, functional status and quality of life, alexithymia, kinesiophobia, catastrophic pain, back awareness, cognitive function evaluated through Oswestry Disability Index(ODI), Nottingham Health Profile (NHP), Toronto Alexithymia Scale, Fear Avoidance Beliefs Questionnaire, Pain Catastrophizing Scale, Fremantle Back Awareness Scale, Montreal Cognitive Assessment respectively. Assessments were repeated before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific low back pain
* Must be pain at least 3 months

Exclusion Criteria:

* History of any lumbar spine surgery
* Presence of neurological deficit
* Having been diagnosed with cardiovascular or systemic diseases that would prevent him / her from taking exercise training.
* The presence of persistent severe pain
* Pain below the knee
* Severe/progressive scoliosis
* Spinal stenosis
* Spondylolisthesis
* Cancer
* Diabetes
* Metabolic syndrome
* Inflammatory, infectious or tumoral disease of the vertebra

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in pain severity | change from baseline in pain severity at 8 weeks
  Patients' average resting, activity and night pain intensities assessed by Visual Analog Scale. The visual analog scale is an 11-point scale ranging from 0 to 10, in which 0 defines absence of pain and 10 describes unbearable pain. Participants asked to rate the average pain levels a horizontal 10 cm straight line on a white sheet from, before and after treatment.
Changes of functional status | change from baseline in functional status at 8 weeks
  Patient's permanent functional disability measured by Oswestry Disability Index. The scale is considered the 'gold standard' of low back functional outcome tools. This scale contain questions related to functional activities of pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling.Interpretation of scale are 0% to 20% for minimal disability, 21% to 40% for moderate disability, 41 % to 60 % for severe disability 61% to 80 % for crippled and 81 % to 100 % Bed-bound.

SECONDARY OUTCOMES:
Changes in quality of life | Change from baseline in life quality levels at 8 weeks
  Health-related quality of life assessed by Nottingham Health Profile (NHP). The NHP contain 38 questions in 6 subareas: pain, physical abilities, energy level, sleep, social isolation and emotional reaction. The scores range from 0 to 100, with each question assigned a weighted value; the sum of all weighted values in a given subarea adds up to 100. Lower scores denoting a better quality of life.
Changes in gait parameters | Change from baseline in gait parameters at 8 weeks
  Gait assessment will be recorded with OptoGait for one minute while participants walked their preferred speed on the treadmill. Patients asked to walk on level surface. Assessment were recorded during one minute.
Changes in metabolic capacity | Change from baseline in metabolic capacity at 8 weeks
  Metabolic capacity testing will be performed according to the Modified Bruce protocol on the Treadmill. At 3 minute intervals, the inclination increase by %2 with a concomitant increase in speed.
Changes in cognitive level | Change from baseline in cognitive level at 8 weeks
  The Montreal Cognitive Assessment Questionnaire (MoCA) will be used to assess the cognitive levels of individuals. MoCA was developed as a rapid screening test for mild cognitive impairment. MoCA assesses various cognitive functions such as attention and concentration, creative functions, memory, language, visual structuring skills, abstract thinking, computation and orientation. The application of MoCA takes about 10 minutes. The maximum total score of the test is 30. A score of 21 or above is considered normal.
Changes in alexithymia | Change from baseline in alexithymia at 8 weeks
  The alexithymia will be assessed by the Toronto Alexithymia Scale (TAS). The scale is a Likert-type self-assessment scale consisting of 20 items and scored between 1-5. Difficulties in recognizing emotions (TAS-1), difficulty in speaking emotions (TAS-2), extroverted thinking (TAS-3) subscales. The individual is asked to select the best option for each item from "Never", "Rarely", "Sometimes", "Often" and "Always". The higher the score, the higher the level of alexithymia.
Changes in kinesiophobia. | Change from baseline in kinesiophobia at 8 weeks
  Fear-Avoidance-Beliefs Questionnaire will be applied to evaluate kinesiophobia which is fear of movement due to low back pain.This questionnaire has 2 sub-sections related to physical activity and work. There are 4 questions scored in the physical activity section and 7 questions in the work section. 0-6 points are obtained for each question. The total score will be recorded. The higher the score, the higher the kinesiophobia.
Changes in back awareness | Change from baseline in back awareness at 8 weeks
  The Fremantle Back Awareness Questionnaire will be used to evaluate how individuals perceive the back according to their body. The questionnaire includes 9 questions that measure how individuals perceive their back according to their body and how they perceive their body position. Questions is answered Likert type as "0" I never feel like this, "4" always or often feel like this.

CONTACTS AND LOCATIONS:
Overall Officials: Müzeyyen ÖZ, MSc, Principal Investigator — Hacettepe University; Özlem Ülger, Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meng XG, Yue SW. Efficacy of aerobic exercise for treatment of chronic low back pain: a meta-analysis. Am J Phys Med Rehabil. 2015 May;94(5):358-65. doi: 10.1097/PHM.0000000000000188. PMID 25299528
- [Background] Inani SB, Selkar SP. Effect of core stabilization exercises versus conventional exercises on pain and functional status in patients with non-specific low back pain: a randomized clinical trial. J Back Musculoskelet Rehabil. 2013;26(1):37-43. doi: 10.3233/BMR-2012-0348. PMID 23411647
- [Background] Chang DG, Holt JA, Sklar M, Groessl EJ. Yoga as a treatment for chronic low back pain: A systematic review of the literature. J Orthop Rheumatol. 2016 Jan 1;3(1):1-8. PMID 27231715
- [Background] Koldas Dogan S, Sonel Tur B, Kurtais Y, Atay MB. Comparison of three different approaches in the treatment of chronic low back pain. Clin Rheumatol. 2008 Jul;27(7):873-81. doi: 10.1007/s10067-007-0815-7. Epub 2008 Jan 11. PMID 18188660